CLINICAL TRIAL: NCT05170906
Title: Cerebral Oxygenation During Vojta Therapy in Healthy Adults Using Near-infrared Spectroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Juan Luis Sanchez Gonzalez, Dr. Juan Luis Sánchez González, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: VojaNeurousal
Record Dates: First submitted 2021-12-11; First posted 2021-12-28 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Healthy; Brain
Keywords: Adult; Vojta Therapy; Oxigenation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The subject will be placed on a stretcher with the torso uncovered. Once the spectroscopy helmet is in place, a recording of the resting activity will be started, two minutes of stimulation (digital pressure), one minute of rest, two minutes of stimulation on the contralateral side and, finally, one minute of rest.
  The therapy consists of the application of a stimulating pressure on the pectoral area in the pattern of the reflex swing locomotion complex in its first phase. For this, the subject will be placed in supine decubitus aligned with respect to the axial axis, with the arms alongside the body, the lower extremities in extension and the head extended with a rotation of approximately 30º to one side of the stimulation. Manual stimulation pressure will be exerted in the space between the 6th-7th or 7th-8th ribs below the mammary line, with a force of about 2 kg.
  Interventions: Other: Reflex locomotion stimulus
- Control Group (Sham Comparator): The subject will be placed on a stretcher with the torso uncovered. Once the adhesive electrodes have been placed in the different recording areas on the anterior part of the trunk, a recording of the activity at rest will begin, two minutes of stimulation (digital pressure), one minute of rest, two minutes of stimulation in the contralateral side and, finally, one minute of rest.
  The control group will receive an application in an area with low receptor density located on the thigh, with a force of about 2 kg
  Interventions: Other: sham stimulus

INTERVENTIONS:
Other: Reflex locomotion stimulus — The therapy consists of the application of a stimulating pressure in the pectoral area in the pattern of the locomotion complex of reflex rolling in its first phase. For this, the subject will be placed in a supine position aligned with respect to the axial axis, with the arms along the body, the lower extremities in extension, and the head extended with a rotation of approximately 30º towards one side of the stimulation. The manual stimulation pressure will be exerted in the space between the 6th-7th or the 7th-8th rib under the mammillary line, with a force of about 2 kg.
  Arms: Experimental Group
Other: sham stimulus — The control group will receive an application in an area with low receptor density located on the thigh, with a force of about 2 kg.
  Arms: Control Group

SUMMARY:
A randomized clinical trial on a cohort of healthy subjects of legal age, both sexes, recruited from the university community and who will be randomly distributed into two groups (experimental and control).

The objective is to assess neurophysiological activation by measuring oxygenation in the supplementary motor and premotor areas of oxygenation in the supplementary motor and premotor areas, through near infrared spectroscopy (NIRS) in healthy subjects spectroscopy (NIRS) in healthy subjects during the application of Vojta Therapy.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old.
* Under 40 years old.
* Full cognitive capacity.

Exclusion Criteria:

* Subjects with neuro-muscular pathologies that affect the abdominal muscles, previous surgeries in the area or any chronic neurological or organic disorder that may alter the results.
* Vaccinated in the 10 days prior to the intervention
* Fever

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Near Infrared Spectroscopy (NIRS) | 15 minutes per patients
  NIRS power

CONTACTS AND LOCATIONS:
Locations (1):
- Juan Luis Sánchez González, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No